CLINICAL TRIAL: NCT04447469
Title: A Phase 2/3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Mavrilimumab (KPL-301) Treatment in Adult Subjects Hospitalized With Severe COVID-19 Pneumonia and Hyper-inflammation
Brief Title: Study of Mavrilimumab (KPL-301) in Participants Hospitalized With Severe Corona Virus Disease 2019 (COVID-19) Pneumonia and Hyper-inflammation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals International, plc (Industry)
Collaborators: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KPL-301-C203
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: COVID
Keywords: COVID-19; pneumonia; hyper-inflammation
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 10 mg/kg (Cohort 1) (Active Comparator): Non-mechanically ventilated participants administered mavrilimumab 10 mg/kg as a single IV infusion
  Interventions: Drug: mavrilimumab
- 6 mg/kg (Cohort 1) (Active Comparator): Non-mechanically ventilated participants administered mavrilimumab 6 mg/kg as a single IV infusion
  Interventions: Drug: mavrilimumab
- Placebo (Cohort 1) (Placebo Comparator): Non-mechanically ventilated participants administered placebo as a single IV infusion
  Interventions: Other: Placebo
- 10 mg/kg (Cohort 2) (Active Comparator): Mechanically ventilated participants administered mavrilimumab 10 mg/kg as a single IV infusion
  Interventions: Drug: mavrilimumab
- 6 mg/kg (Cohort 2) (Active Comparator): Mechanically ventilated participants administered mavrilimumab 6 mg/kg as a single IV infusion
  Interventions: Drug: mavrilimumab
- Placebo (Cohort 2) (Placebo Comparator): Mechanically ventilated participants administered placebo as a single IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: mavrilimumab — anti-granulocyte-macrophage colony-stimulating factor receptor alpha (GM-CSF-Rα) monoclonal antibody (human isoform immunoglobulin G [IgG4])
  Other Names: KPL-301; CAM3001
  Arms: 10 mg/kg (Cohort 1); 10 mg/kg (Cohort 2); 6 mg/kg (Cohort 1); 6 mg/kg (Cohort 2)
Other: Placebo — matching placebo
  Arms: Placebo (Cohort 1); Placebo (Cohort 2)

SUMMARY:
Interventional, randomized, double-blind, placebo-controlled study encompassing 2 development phases (Phase 2 and Phase 3).

DETAILED DESCRIPTION:
The Phase 2 portion of the study will evaluate the efficacy and safety of 2 dose levels of mavrilimumab relative to placebo (standard of care) in participants who have tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) with x-ray/computed tomography (CT) evidence of bilateral pneumonia and active or recent signs of hyperinflammation (fever or clinical laboratory results indicative of hyper-inflammation). The Phase 3 portion is intended to confirm Phase 2 efficacy and safety findings. In both Phase 2 and Phase 3, participants will be enrolled into 2 cohorts: Cohort 1 will include non-mechanically ventilated, hospitalized participants who require supplemental oxygen to maintain oxygen saturation (SpO2) ≥ 92% (ie, "non-mechanically ventilated" participants); Cohort 2 will include hospitalized participants for whom mechanical ventilation was recently initiated (ie, "mechanically ventilated" participants). Following Screening, enrolled participants in each cohort will be randomized 1:1:1 to receive one of 2 mavrilimumab dose levels, or placebo as a single intravenous (IV) infusion (Day 1). Participants will undergo primary study assessments through Day 29 and will be followed for safety through Day 90.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject (or legally authorized representative) is able and willing to provide informed consent, which includes compliance with study requirements and restrictions listed in the consent form. Consent must be performed per institutional regulations.
* Age of ≥ 18 years
* Positive SARS-CoV-2 (2019-nCoV) test within 14 days prior to randomization
* Hospitalized for SARS-CoV-2 (2019-nCoV)
* Bilateral pneumonia on chest x-ray or computed tomography
* Clinical laboratory results indicative of hyper-inflammation within 7 days prior to randomization
* Cohort 1: Receiving any form of non-invasive ventilation OR oxygenation to maintain SpO2 ≥ 92% and non-mechanically ventilated (examples include nasal cannula, face mask, venturi mask, high-flow nasal cannula, or non-invasive positive pressure ventilation)
* Cohort 2: Recently ventilated with mechanical ventilation beginning within 48 hours prior to randomization

Key Exclusion Criteria:

* Onset of COVID-19 symptoms > 14 days prior to randomization
* Hospitalized > 7 days prior to randomization
* Need for invasive mechanical ventilation (Only for Cohort 1)
* Need for ECMO
* Serious prior or concomitant illness that in the opinion of the Investigator precludes the subject from enrolling in the trial
* Recent treatment with cell-depleting biological therapies (eg, anti-CD20) within 12 months, non-cell-depleting biological therapies (such as anti-tumor necrosis factor [TNF], anakinra, anti-IL-6 receptor [eg, tocilizumab], or abatacept) within 8 weeks (or 5 half-lives, whichever is longer), treatment with alkylating agents within 12 weeks, treatment with cyclosporine A, azathioprine, cyclophosphamide, mycophenolate mofetil (MMF), or other immunosuppressant (except for corticosteroids) within 4 weeks prior to randomization. Medications that become standard of care for COVID-19 and/or receive emergency use authorization may be allowed after discussion with the medical monitor.
* If subject is receiving or has received hydroxychloroquine within 3 months prior to screening visit, a corrected QT interval by Federicia method (QTcF) on Screening electrocardiogram (ECG) ≥500ms is exclusionary. If subject has a pacemaker, this criterion does not apply.
* Enrolled in another investigational study of a medical intervention within 30 days prior to randomization. Participation in open label trials involving investigational treatments for COVID-19 may be allowed upon approval by the Sponsor.
* Life expectancy less than 48 hours, in the opinion of the Investigator
* Known human immunodeficiency virus infection (regardless of immunological status), known hepatitis B virus surface antigen positivity and/or anti-hepatitis C virus positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (9):
  - UCLA Medical Center, Los Angeles, California
  - SHARP Health Care, San Diego, California
  - Affinity Health, Chicago, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Allina Health System, Minneapolis, Minnesota
  - Mercy Clinic Hospitalists, Springfield, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - University of Texas Health Sciences, Houston, Texas
- Brazil (11):
  - Hospital Cardio Pulmonar, Salvador, Estado de Bahia
  - Hospital Luxemburgo - Associação Mário Penna, Belo Horizonte, Minas Gerais
  - CPCLIN - Centro de Pesquisas Clínicas, Natal, Rio Grande do Norte
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - UPECLIN - Unidade de Pesquisa Clínica, Botucatu, São Paulo
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Hospital Adventista de Belem, Belém
  - IEP HGF - Instituto de Estudos e Pesquisas Clinicas do Ceará, Fortaleza
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José
  - Hospital Alemão Oswaldo Cruz, São Paulo
- Chile (2):
  - Clinica Las Condes, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
- Peru (4):
  - Hospital Nacional Alberto Sabogal Sologuren, Bellavista
  - Essalud - Hospital de Emergencias Grau, Lima Cercado
  - Hospital Nacional Cayetano Heredia, San Martín de Porres
  - Clinica Providencia, San Miguel
- South Africa (6):
  - University of Cape Town - Lung Institute, Cape Town, Western Cape
  - IATROS International, Bloemfontein
  - Tiervlei Trial Center, Cape Town
  - TASK Eden, George
  - Into Research - Little Company of Mary Medical Center, Pretoria
  - Limpopo Clinical Research Initiative, Rustenburg

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will review IPD requests proposals from qualified researchers
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests will be accepted after publication of the primary data manuscript
Access Criteria: IPD access will be provided to qualified academic researchers pending the Sponsor's review of the proposed research, including scientific novelty, review of the analytical and publication plans, funding source of the proposed research, any potential conflicts of interest, and institutional capabilities to perform the planned research.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were divided into 2 cohorts (non-mechanically ventilated and mechanically ventilated) and randomized 1:1:1 to receive a single IV infusion of mavrilimumab (10 mg/kg or 6 mg/kg) or placebo in addition to standard of care. There was a seamless transition in enrollment in both cohorts between the Phase 2 and Phase 3 portions of the study. (For each cohort, once the last participant in Phase 2 was enrolled, all subsequent participants were considered Phase 3 participants.)
Groups:
- Phase 2: 10 mg/kg (Cohort 1); Phase 3: 10 mg/kg (Cohort 1): Non-mechanically ventilated participants administered mavrilimumab 10 mg/kg as a single IV infusion
- Phase 2: 6 mg/kg (Cohort 1); Phase 3: 6 mg/kg (Cohort 1): Non-mechanically ventilated participants administered mavrilimumab 6 mg/kg as a single IV infusion
- Phase 2: Placebo (Cohort 1); Phase 3: Placebo (Cohort 1): Non-mechanically ventilated participants administered placebo as a single IV infusion
- Phase 2: 10 mg/kg (Cohort 2); Phase 3: 10 mg/kg (Cohort 2): Mechanically ventilated participants administered mavrilimumab 10 mg/kg as a single IV infusion
- Phase 2: 6 mg/kg (Cohort 2); Phase 3: 6 mg/kg (Cohort 2): Mechanically ventilated participants administered mavrilimumab 6 mg/kg as a single IV infusion
- Phase 2: Placebo (Cohort 2); Phase 3: Placebo (Cohort 2): Mechanically ventilated participants administered placebo as a single IV infusion
Period: Overall Study
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1) | Phase 2: 10 mg/kg (Cohort 2) | Phase 2: 6 mg/kg (Cohort 2) | Phase 2: Placebo (Cohort 2) | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1) | Phase 3: 10 mg/kg (Cohort 2) | Phase 3: 6 mg/kg (Cohort 2) | Phase 3: Placebo (Cohort 2)
Started (Enrolled) | 37 | 42 | 41 | 18 | 15 | 17 | 198 | 192 | 192 | 20 | 22 | 20
Enrolled and Treated | 35 | 41 | 40 | 15 | 15 | 17 | 195 | 188 | 191 | 20 | 21 | 20
Completed | 29 | 32 | 28 | 7 | 6 | 7 | 162 | 154 | 150 | 9 | 12 | 7
Not Completed | 8 | 10 | 13 | 11 | 9 | 10 | 36 | 38 | 42 | 11 | 10 | 13

BASELINE CHARACTERISTICS:
Population: Phase 2: Modified Intent-to-Treat (mITT) Analysis Set: All randomized participants who passed screening and received study drug (two enrolled and treated participants [1 each in the 6 mg/kg and placebo groups] were randomized and dosed in violation of inclusion/exclusion criteria and were thus excluded from this Set); Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1) | Phase 2: 10 mg/kg (Cohort 2) | Phase 2: 6 mg/kg (Cohort 2) | Phase 2: Placebo (Cohort 2) | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1) | Phase 3: 10 mg/kg (Cohort 2) | Phase 3: 6 mg/kg (Cohort 2) | Phase 3: Placebo (Cohort 2) | Total
Number analyzed (Participants) | 35 | 40 | 39 | 15 | 15 | 17 | 198 | 192 | 192 | 20 | 22 | 20 | 805
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.89) | 56.9 (14.36) | 57.4 (14.29) | 61.1 (11.54) | 59.3 (15.89) | 56.9 (15.14) | 52.5 (14.03) | 51.3 (14.32) | 52.2 (14.00) | 59.2 (14.65) | 57.2 (13.20) | 55.80 (14.75) | 53.55 (14.29)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 24 | 30 | 27 | 10 | 9 | 11 | 159 | 157 | 155 | 13 | 14 | 14 | 623
  ≥ 65 years | 11 | 10 | 12 | 5 | 6 | 6 | 39 | 35 | 37 | 7 | 8 | 6 | 182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 18 | 3 | 4 | 6 | 66 | 66 | 66 | 9 | 5 | 7 | 281
  Male | 23 | 21 | 21 | 12 | 11 | 11 | 132 | 126 | 126 | 11 | 17 | 13 | 524
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 11 | 9 | 4 | 8 | 122 | 107 | 118 | 13 | 17 | 16 | 447
  Not Hispanic or Latino | 18 | 21 | 20 | 4 | 9 | 7 | 38 | 37 | 33 | 2 | 1 | 2 | 192
  Unknown or Not Reported | 5 | 9 | 8 | 2 | 2 | 2 | 38 | 48 | 41 | 5 | 4 | 2 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 1 | 1 | 3 | 9 | 4 | 1 | 0 | 0 | 22
  Asian | 0 | 1 | 2 | 1 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 4 | 3 | 2 | 2 | 15 | 16 | 11 | 0 | 1 | 1 | 66
  White | 19 | 25 | 21 | 9 | 7 | 11 | 142 | 134 | 143 | 15 | 13 | 16 | 555
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 6
  Unknown or Not Reported | 8 | 8 | 11 | 2 | 5 | 3 | 33 | 30 | 31 | 4 | 8 | 3 | 146
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 12 | 15 | 4 | 4 | 5 | 25 | 23 | 20 | 0 | 0 | 0 | 117
  Brazil | 14 | 18 | 11 | 10 | 5 | 6 | 153 | 143 | 150 | 16 | 19 | 17 | 562
  South Africa | 9 | 10 | 12 | 1 | 5 | 4 | 13 | 15 | 16 | 1 | 1 | 2 | 89
  Chile | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 1 | 1 | 11
  Peru | 2 | 0 | 1 | 0 | 1 | 2 | 4 | 8 | 5 | 2 | 1 | 0 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1, Phase 2: Percentage of Participants Alive and Free of Mechanical Ventilation at Day 29
Description: Mechanical ventilation is defined as invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO). Mechanical ventilation status was evaluated based on the National Institute of Allergy and Infectious Diseases (NIAID) clinical outcome 8-point ordinal scale. Participants whose clinical outcome met a NIAID score of 2 were considered as using mechanical ventilation.
  The NIAID score is an 8-point ordinal scale of clinical outcomes: 1=death; 2=hospitalized, on invasive mechanical ventilation or ECMO; 3=hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5=hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID 19 related or otherwise); 6=hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7=not hospitalized, limitation on activities and/or requiring home oxygen; 8=not hospitalized, no limitations on activities.
Time Frame: Day 29
Population: Phase 2: Modified Intent-to-Treat (mITT) Analysis Set: All randomized participants who passed screening and received study drug (two enrolled and treated participants [1 each in the 6 mg/kg and placebo groups] were randomized and dosed in violation of inclusion/exclusion criteria and were thus excluded from this Set).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1)
Number analyzed (Participants) | 35 | 40 | 39
percentage of participants | 85.7 [69.7 to 95.2] | 87.5 [73.2 to 95.8] | 74.4 [57.9 to 87.0]
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.2598, Fisher Exact — P-value and odds ratio were calculated using Fisher's Exact test; Odds Ratio (OR) = 2.069, 95% CI 2-sided [0.555 to 8.615]
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.1610, Fisher Exact — P-value and odds ratio were calculated using Fisher's Exact test; Odds Ratio (OR) = 2.414, 95% CI 2-sided [0.653 to 9.957]
Statistical Analysis 3: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.2448, Cochran-Mantel-Haenszel — P-value and odds ratio were calculated using Cochran Mantel-Haenszel (CMH) test, stratified by randomization strata (standard of care antiretroviral therapy, age, and ARDS status); Stratified Odds Ratio = 2.091, 95% CI 2-sided [0.612 to 7.144]
Statistical Analysis 4: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.1378, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]; Stratified Odds Ratio = 2.749, 95% CI 2-sided [0.756 to 9.993]

2. Primary Outcome: Cohort 1, Phase 3: Percentage of Participants Alive and Free of Mechanical Ventilation at Day 29
Description: as for outcome 1
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1)
Number analyzed (Participants) | 198 | 192 | 192
percentage of participants | 84.3 [78.5 to 89.1] | 82.8 [76.7 to 87.9] | 81.3 [75.0 to 86.5]
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.4534, Cochran-Mantel-Haenszel — P-value and odds ratio were calculated using Cochran Mantel-Haenszel (CMH) test, stratified by randomization strata (age and ARDS status); Stratified Odds Ratio = 1.231, 95% CI 2-sided [0.715 to 2.120]
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.7414, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Stratified Odds Ratio = 1.097, 95% CI 2-sided [0.636 to 1.891]

3. Primary Outcome: Cohort 2, Phase 2: Percentage of Participants Who Died by Day 29
Description: Defined as the proportion of subjects with mechanical ventilation who have died by Day 29.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 10 mg/kg (Cohort 2) | Phase 2: 6 mg/kg (Cohort 2) | Phase 2: Placebo (Cohort 2)
Number analyzed (Participants) | 15 | 15 | 17
percentage of participants | 46.7 [21.3 to 73.4] | 53.3 [26.6 to 78.7] | 47.1 [23.0 to 72.2]
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 2) vs Phase 2: Placebo (Cohort 2); Test type: Superiority; p = 1.0000, Fisher Exact; Odds Ratio (OR) = 0.984, 95% CI 2-sided [0.198 to 4.884]
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 2) vs Phase 2: Placebo (Cohort 2); Test type: Superiority; p = 1.0000, Fisher Exact; Odds Ratio (OR) = 1.286, 95% CI 2-sided [0.260 to 6.417]

4. Primary Outcome: Cohort 2, Phase 3: Percentage of Participants Who Died by Day 29
Description: Defined as the proportion of subjects with mechanical ventilation who have died by Day 29.
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: 10 mg/kg (Cohort 2) | Phase 3: 6 mg/kg (Cohort 2) | Phase 3: Placebo (Cohort 2)
Number analyzed (Participants) | 20 | 22 | 20
percentage of participants | 40.0 [19.1 to 63.9] | 27.3 [10.7 to 50.2] | 55.0 [31.5 to 76.9]
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 2) vs Phase 3: Placebo (Cohort 2); Test type: Superiority; Difference in Proportion = -15.0, 95% CI 2-sided [-45.6 to 15.6] — 95% CI were calculated using asymptotic normal approximation. Difference = KPL-301 - placebo
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 2) vs Phase 3: Placebo (Cohort 2); Test type: Superiority; Difference in Proportions = -27.7, 95% CI 2-sided [-56.4 to 0.9] — 95% CI were calculated using asymptotic normal approximation. Difference = KPL-301 - Placebo

5. Secondary Outcome: Cohort 1, Phase 2: Time to 2-point Clinical Improvement by Day 29
Description: Defined as time from randomization to a 2-point improvement on the NIAID 8-point ordinal scale, or discharge from the hospital, whichever came first. Participants who died before Day 29 were censored at Day 30. Kaplan-Meier method used to estimate the survival functions for each treatment arm.
  The NIAID score is an 8-point ordinal scale of clinical outcomes: 1=death; 2=hospitalized, on invasive mechanical ventilation or ECMO; 3=hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5=hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID 19 related or otherwise); 6=hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7=not hospitalized, limitation on activities and/or requiring home oxygen; 8=not hospitalized, no limitations on activities.
Time Frame: Day 29
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1)
Number analyzed (Participants) | 35 | 40 | 39
days | 8.0 [6.0 to 8.0] | 7.0 [7.0 to 8.0] | 11.0 [6.0 to 14.0]
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.6229, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, age, and ARDS status)
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.5526, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, age, and ARDS status)

6. Secondary Outcome: Phase 2, Cohort 1: Time to Return to Room Air or Discharge by Day 29
Description: Defined as time from randomization to breathing room air (NIAID score ≥ 5), or discharge from the hospital, whichever came first. Participants who died before Day 29 were censored at Day 30.
Time Frame: Day 29
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1)
Number analyzed (Participants) | 35 | 40 | 39
days | 7.0 [6.0 to 8.0] | 7.0 [6.0 to 7.0] | 9.0 [6.0 to 13.0]
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.9426, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, age, and ARDS status); Hazard Ratio (HR) = 1.02, 80% CI 2-sided [0.71 to 1.46] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata (Standard of Care antiretroviral therapy, age, and ARDS status)
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.6838, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, age, and ARDS status); Hazard Ratio (HR) = 1.11, 80% CI 2-sided [0.78 to 1.57] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Phase 2, Cohort 1: Percentage of Participants Who Die by Day 29
Description: 95% CI were calculated using Clopper-Pearson exact method based on the beta distribution.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1)
Number analyzed (Participants) | 35 | 40 | 39
percentage of participants | 5.7 [0.7 to 19.2] | 10.0 [2.8 to 23.7] | 20.5 [9.3 to 36.5]
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.0905, Fisher Exact; Odds Ratio (OR) = 0.235, 95% CI 2-sided [0.023 to 1.328]
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.2247, Fisher Exact; Odds Ratio (OR) = 0.431, 95% CI 2-sided [0.087 to 1.815]
Statistical Analysis 3: Comparison: Phase 2: 10 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.0623, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]; Stratified Odds Ratio = 0.191, 95% CI 2-sided [0.033 to 1.114]
Statistical Analysis 4: Comparison: Phase 2: 6 mg/kg (Cohort 1) vs Phase 2: Placebo (Cohort 1); Test type: Superiority; p = 0.1957, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 3]; Stratified Odds Ratio = 0.368, 95% CI 2-sided [0.085 to 1.583]

8. Secondary Outcome: Phase 2, Cohort 2: Time to 1-Point Clinical Improvement by Day 29
Description: Defined as time from randomization to the date of a 1-point improvement on the NIAID score 8-point ordinal scale or discharge from the hospital, whichever occurred first, by Day 29. Participants who did not have 1-point improvement on the NIAID nor discharge from the hospital were censored at the date of the last NIAID 8-point ordinal scale assessment on/before Day 29. Participants who died were censored at Day 32.
Time Frame: Day 29
Population: Phase 2: Modified Intent-to-Treat (mITT) Analysis Set: All randomized participants who passed screening and received study drug.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Phase 2: 10 mg/kg (Cohort 2) | Phase 2: 6 mg/kg (Cohort 2) | Phase 2: Placebo (Cohort 2)
Number analyzed (Participants) | 15 | 15 | 17
days | 28.0 [16.0 to NA] — Median and upper CI were not estimable using Kaplan-Meier method due to insufficient number of participants with events | NA [19.0 to NA] — Median and upper CI were not estimable using Kaplan-Meier method due to insufficient number of participants with events | NA [16.0 to NA] — Median and upper CI were not estimable using Kaplan-Meier method due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Phase 2: 10 mg/kg (Cohort 2) vs Phase 2: Placebo (Cohort 2); Test type: Superiority; p = 0.3766, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, and age); Hazard Ratio (HR) = 1.57, 80% CI 2-sided [0.80 to 3.09] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata (Standard of Care antiretroviral therapy and age)
Statistical Analysis 2: Comparison: Phase 2: 6 mg/kg (Cohort 2) vs Phase 2: Placebo (Cohort 2); Test type: Superiority; p = 0.9209, Log Rank — Log-rank test is stratified by randomization strata (Standard of Care antiretroviral therapy, and age); Hazard Ratio (HR) = 1.05, 80% CI 2-sided [0.51 to 2.16] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Phase 3, Cohort 1: Percentage of Participants Who Died at Day 29
Description: Mortality rate at day 29 is the proportion of subjects who die by day 29. 95% CI were calculated using Clopper-Pearson exact method based on the beta distribution.
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1)
Number analyzed (Participants) | 198 | 192 | 192
percentage of participants | 9.6 [5.9 to 14.6] | 14.1 [9.5 to 19.8] | 14.1 [9.5 to 19.8]
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.1772, Cochran-Mantel-Haenszel — Calculated using Cochran Mantel-Haenszel test, stratified by randomization strata (age and ARDS status); Stratified Odds Ratio = 0.645, 95% CI 2-sided [0.340 to 1.222]
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.9269, Cochran-Mantel-Haenszel — Calculated using Cochran Mantel-Haenszel test, stratified by randomization strata (age and ARDS status); Stratified Odds Ratio = 1.029, 95% CI 2-sided [0.563 to 1.881]

10. Secondary Outcome: Phase 3, Cohort 1: Ventilation-Free Survival (Time to Ventilation or Death) by Day 29
Description: Time to ventilation or death by Day 29 was defined as time (in days) from randomization to the date of death or start date of using mechanical ventilation (NIAID score ≤ 2) by Day 29. Participants who never had NIAID score ≤ 2 by Day 29 were censored at last assessment date of NIAID 8-point ordinal scale.
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1)
Number analyzed (Participants) | 198 | 192 | 192
days | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.9578, Log Rank — Log-rank test is stratified by randomization strata (age, and ARDS status); Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.66 to 1.49] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata (age and ARDS status)
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.5274, Log Rank — Log-rank test is stratified by randomization strata (age, and ARDS status); Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.76 to 1.70] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Phase 3, Cohort 1: Overall Survival by Day 29
Description: Overall survival was defined as time from randomization to the date of death on/before Day 29. Participants who did not have a death record by Day 29 were censored at last date known alive on/before Day 29.
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1)
Number analyzed (Participants) | 198 | 192 | 192
days | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events | NA [NA to NA] — Not estimable using the Kaplan-Meier method due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.1336, Log Rank — Log-rank test is stratified by randomization strata (age, and ARDS status); Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.36 to 1.15] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata (age, and ARDS status)
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 1) vs Phase 3: Placebo (Cohort 1); Test type: Superiority; p = 0.9767, Log Rank — Log-rank test is stratified by randomization strata (age, and ARDS status); Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.59 to 1.72] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata ( age, and ARDS status)

12. Secondary Outcome: Phase 3, Cohort 2: Time to 1-point Clinical Improvement by Day 29
Description: Defined as time from randomization to the date of a 1-point improvement on the NIAID 8-point ordinal scale or discharge from the hospital, whichever occurred first, by Day 29. Participants who did not have 1-point improvement on the NIAID nor discharge from the hospital were censored at the date of the last NIAID 8-point ordinal scale assessment on/before Day 29. Participants who died were censored at Day 35.
Time Frame: Day 29
Population: Phase 3: Intent-to-Treat (ITT) Analysis Set: All randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3: 10 mg/kg (Cohort 2) | Phase 3: 6 mg/kg (Cohort 2) | Phase 3: Placebo (Cohort 2)
Number analyzed (Participants) | 20 | 22 | 20
days | NA [9.0 to NA] — Median and upper limit confidence interval were not estimable using Kaplan-Meier method due to insufficient number of participants with events | 21.5 [8.0 to NA] — Upper limit confidence interval was not estimable using Kaplan-Meier method due to insufficient number of participants with events | NA [12.0 to NA] — Median and upper limit confidence interval were not estimable using Kaplan-Meier method due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Phase 3: 10 mg/kg (Cohort 2) vs Phase 3: Placebo (Cohort 2); Test type: Superiority; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.55 to 3.71] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by randomization strata (age)
Statistical Analysis 2: Comparison: Phase 3: 6 mg/kg (Cohort 2) vs Phase 3: Placebo (Cohort 2); Test type: Superiority; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [0.78 to 4.54] — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: From enrollment (all-cause mortality) or first dose of study drug (adverse events) to the end of study; the maximum study duration was 44 weeks.
Arm/Group | Phase 2: 10 mg/kg (Cohort 1) | Phase 2: 6 mg/kg (Cohort 1) | Phase 2: Placebo (Cohort 1) | Phase 2: 10 mg/kg (Cohort 2) | Phase 2: 6 mg/kg (Cohort 2) | Phase 2: Placebo (Cohort 2) | Phase 3: 10 mg/kg (Cohort 1) | Phase 3: 6 mg/kg (Cohort 1) | Phase 3: Placebo (Cohort 1) | Phase 3: 10 mg/kg (Cohort 2) | Phase 3: 6 mg/kg (Cohort 2) | Phase 3: Placebo (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 4/35 | 5/41 | 9/40 | 7/15 | 9/15 | 9/17 | 20/195 | 30/188 | 30/191 | 7/20 | 8/21 | 12/20
Serious Adverse Events (participants affected / at risk) | 5/35 | 7/41 | 13/40 | 10/15 | 12/15 | 10/17 | 48/195 | 49/188 | 43/191 | 13/20 | 14/21 | 15/20
Other Adverse Events (participants affected / at risk) | 19/35 | 18/41 | 23/40 | 11/15 | 12/15 | 14/17 | 90/195 | 86/188 | 83/191 | 12/20 | 13/21 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: 10 mg/kg (Cohort 1) (N=35) | Phase 2: 6 mg/kg (Cohort 1) (N=41) | Phase 2: Placebo (Cohort 1) (N=40) | Phase 2: 10 mg/kg (Cohort 2) (N=15) | Phase 2: 6 mg/kg (Cohort 2) (N=15) | Phase 2: Placebo (Cohort 2) (N=17) | Phase 3: 10 mg/kg (Cohort 1) (N=195) | Phase 3: 6 mg/kg (Cohort 1) (N=188) | Phase 3: Placebo (Cohort 1) (N=191) | Phase 3: 10 mg/kg (Cohort 2) (N=20) | Phase 3: 6 mg/kg (Cohort 2) (N=21) | Phase 3: Placebo (Cohort 2) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pituitary apoplexy (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Brain death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site haemorrhage (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 5 | 6 | 2 | 2 | 4
Pneumonia acinetobacter (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 4 | 3 | 1 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 8 | 9 | 7 | 0 | 0 | 4
Septic shock (Infections and infestations) | 0 | 2 | 4 | 0 | 2 | 4 | 10 | 13 | 15 | 3 | 2 | 7
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Severe acute respiratory syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Tracheobronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Urinary tract candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 1 | 1 | 2 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 8 | 11 | 12 | 1 | 4 | 4
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 4 | 4 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 4 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 9 | 8 | 5 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 4 | 1 | 2 | 4 | 5 | 6 | 1 | 0 | 2
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: 10 mg/kg (Cohort 1) (N=35) | Phase 2: 6 mg/kg (Cohort 1) (N=41) | Phase 2: Placebo (Cohort 1) (N=40) | Phase 2: 10 mg/kg (Cohort 2) (N=15) | Phase 2: 6 mg/kg (Cohort 2) (N=15) | Phase 2: Placebo (Cohort 2) (N=17) | Phase 3: 10 mg/kg (Cohort 1) (N=195) | Phase 3: 6 mg/kg (Cohort 1) (N=188) | Phase 3: Placebo (Cohort 1) (N=191) | Phase 3: 10 mg/kg (Cohort 2) (N=20) | Phase 3: 6 mg/kg (Cohort 2) (N=21) | Phase 3: Placebo (Cohort 2) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 11 | 5 | 5 | 2 | 3 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 5 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Familial tremor (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 1 | 0 | 8 | 8 | 8 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acinetobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acinetobacter sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burkholderia cepacia complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 2 | 6 | 7 | 8 | 2 | 4 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 1 | 4 | 1 | 3 | 2 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Relapsing fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sedation complication (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 2
Tracheobronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 1 | 0 | 1 | 5 | 4 | 2 | 2 | 1 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gram stain positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mean arterial pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulse pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sputum culture positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Strongyloides test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 6 | 6 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 4 | 4 | 1 | 0 | 0 | 0
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 6 | 5 | 1 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 5 | 1 | 1 | 1 | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 1 | 2 | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 5 | 1 | 1 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 12 | 8 | 7 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 3 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meige's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 4 | 2 | 1 | 0 | 1 | 3 | 1 | 4 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 3 | 5 | 1 | 0 | 0 | 0
Intensive care unit delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 6 | 6 | 7 | 2 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 2 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 4 | 3 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 7 | 7 | 7 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 7 | 9 | 2 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 2 | 0
Microangiopathy (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Venous haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or presentation of data related to the Clinical Trial, including but not limited to, publications in specialized journals or disclosures in Medical Congresses, must be previously authorized in writing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT04447469/Prot_SAP_000.pdf